CLINICAL TRIAL: NCT05854056
Title: Effect of Accelerated Postoperative Rehabilitation After Tibial Tubercle Distalisation: a Randomised Controlled Trial Protocol
Brief Title: Tibial Tubercle Distalisation and Accelerated Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Pihlajalinna Hospital, Tampere (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R22072
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Patella Alta; Tibial Tubercle Distalisation Osteotomy; Rehabilitation
Keywords: Patella Alta; Tibial tubercle distalisation osteotomy; Accelerated rehabilitation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accelerated rehabilitation protocol (Active Comparator): Elements of physical therapy Group 1 Accelerated rehabilitation Antioedema knee, calf, leg Day 1 Knee brace, ROM limitations No Weight-bearing limitations No, crutches are recommended for 4 weeks. Active exercises. Functional exercises. 1 week Active dynamic strengthening exercises. 5 weeks Closed chain exercises for muscle strengthening. 8 weeks Muscle endurance and neuromuscular control, progress strengthening exercises, jogging 12 weeks
  Interventions: Procedure: Accelerated rehabilitation protocol
- Conservative rehabilitation protocol (Active Comparator): Elements of physical therapy Group 2 Conservative rehabilitation Antioedema knee, calf, leg Day 1 Knee brace, ROM limitations 6 weeks Weight-bearing limitations 4 weeks limb weight, followed by half body weight till week 6
  Active exercises. Functional exercises. 8 weeks Active dynamic strengthening exercises. 8 weeks Closed chain exercises for muscle strengthening. 8 weeks Muscle endurance and neuromuscular control, progress strengthening exercises, jogging 12 weeks
  Interventions: Procedure: Conservative rehabilitation protocol

INTERVENTIONS:
Procedure: Accelerated rehabilitation protocol — See Arms section
  Arms: Accelerated rehabilitation protocol
Procedure: Conservative rehabilitation protocol — See Arms section
  Arms: Conservative rehabilitation protocol

SUMMARY:
The goal of this clinical trial is to compare in distalising tibial tubercle osteotomy procedure group fast rehabilitation to traditional rehabilitation.

The main questions it aims to answer are:

* Will the novel accelerated rehabilitation protocol lead to faster recovery and improved functional outcome at 6, 12 and 24 weeks compared with the conservative rehabilitation protocol?
* Will the complication rate be similar in both groups?

Participants will be following fast rehabilitation or the traditional rehabilitation guidelines after distalising tibial tubercle osteotomy procedure according to the randomisation.

Researchers will compare fast rehabilitation group to the traditional rehabilitation group to see if recovery and functional outcome is improved in fast rehabilitation group and complication rate will be similar in both groups.

DETAILED DESCRIPTION:
Patella alta is a clinical condition where the patella is positioned too proximal in relation to the femoral trochlea. Such an abnormality may cause patellar instability and predispose to recurrent patellofemoral dislocations and patellofemoral pain. There are no conclusive guidelines for determining a threshold for too high positioned patella, as several different methods have been described to measure patellar height. As a surgical solution, distalising tibial tubercle osteotomy has been described to correct excessive patellar height.

In the early phase of the distalising tibial tubercle osteotomy postoperative protocol, weightbearing and knee flexion are limited with a brace commonly for 4-8 weeks. The potential risks for adverse effects associated with the limitation rehabilitation protocol include a delay in regaining knee range of motion, stiffness and muscle weakness. As a result, recovery from surgery is delayed and may lead to additional procedures and long-term morbidity in knee function.

This is a prospective, randomised, controlled, single-blinded, single centre trial comparing a novel accelerated rehabilitation protocol with the traditional, motion restricting rehabilitation protocol. All skeletally mature patients aged 35 years and younger, referred to as the distalising tibial tubercle osteotomy procedure group, are eligible for inclusion in the study. Patients will be randomised to either the fast rehabilitation group or the traditional rehabilitation group. Patients with patellar instability will be additionally treated with medial patellofemoral ligament reconstruction.

The hypothesis of the trial is that the novel accelerated rehabilitation protocol will lead to faster recovery and improved functional outcome at 6, 12 and 24 weeks compared with the conservative rehabilitation protocol. A secondary hypothesis is that the complication rate will be similar in both groups.

The study will document short-term recovery and the planned follow-up will be 3 years. After the 1-year follow-up, the trial results will be disseminated in a major peer-reviewed orthopaedic publication.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patella alta with recurrent dislocation or subluxation. Long-lasting anterior knee pain not responding to rehabilitation.

Exclusion Criteria:

Radiographic:

* Open growth plates
* Iwano [8] grade III and IV changes in patellofemoral joint
* Caton-Deschamps <1.1 in MRI
* PTI >50% in MRI
* High grade trochlear dysplasia

General:

* Refuses to participate in the study
* Aged less than 15 or more than 35 years
* Severe neurological, pulmonal or cardiovascular comorbidities that are contraindications for surgery
* Lack of adequate co-operation
* Does not adequately understand written and spoken instructions in the local language

Those patients who decline to take part in the trial will be asked to join a follow-up cohort as a background population. The patients in this follow-up cohort will be treated "as normal" without allocation, but the follow-up questionnaires will be the same as those given to the randomly assigned population. The patients in the follow-up cohort will also be asked to provide informed written consent.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome in this study will be knee range of motion (ROM) measured at 12 weeks postoperatively. | At 12 weeks
  A difference of 10º in full range of movement will be considered significant. The results will be measured with a long goniometer in a standardised manner.

SECONDARY OUTCOMES:
Secondary outcomes will be knee the Knee Injury and Osteoarthritis Outcome Score (KOOS). | measured at baseline, 6, 24 and 52 weeks postoperatively
  KOOS consists of 5 subscales: Pain, other Symptoms, Function in daily living, Function in sport and recreation and knee related Quality of life. The baseline score from KOOS is recorded during the physiotherapist visit.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Weitz, Study Chair — Pihlajalinna; Ville M Mattila, Prof, Study Chair — Department of Orthopaedic Surgery, Tampere University Hospital, Tampere, Finland; Erkki Nilkku, Study Chair — Pihlajalinna; Petri J Sillanpää, Study Chair — Pihlajalinna

IPD SHARING:
Plan to Share IPD: No
The copyright of the trial research data will be owned and created by the participating research parties. The data will be shared among all participating researchers who will receive access to the data after the trial is completed. Due to confidentiality and legal agreements, public data sharing will be restricted because we only have permission to hold the data in the specific research server, not to transfer data. Under certain circumstances, for example, when a new member joins the collaboration, we will grant access to the data.

REFERENCES:
- [Background] Biedert RM, Tscholl PM. Patella Alta: A Comprehensive Review of Current Knowledge. Am J Orthop (Belle Mead NJ). 2017 Nov/Dec;46(6):290-300. PMID 29309446
- [Background] Insall J, Salvati E. Patella position in the normal knee joint. Radiology. 1971 Oct;101(1):101-4. doi: 10.1148/101.1.101. No abstract available. PMID 5111961
- [Background] Caton J. [Method of measuring the height of the patella]. Acta Orthop Belg. 1989;55(3):385-6. French. PMID 2603679
- [Background] Caton J, Mironneau A, Walch G, Levigne C, Michel CR. [Idiopathic high patella in adolescents. Apropos of 61 surgical cases]. Rev Chir Orthop Reparatrice Appar Mot. 1990;76(4):253-60. French. PMID 2148403
- [Background] Sherman SL, Erickson BJ, Cvetanovich GL, Chalmers PN, Farr J 2nd, Bach BR Jr, Cole BJ. Tibial Tuberosity Osteotomy: Indications, Techniques, and Outcomes. Am J Sports Med. 2014 Aug;42(8):2006-17. doi: 10.1177/0363546513507423. Epub 2013 Nov 6. PMID 24197613
- [Background] Ambra LF, Phan A, Gomoll AH. A New Technique for Distalization of the Tibial Tubercle That Allows Preservation of the Proximal Buttress. Orthop J Sports Med. 2018 Sep 25;6(9):2325967118798621. doi: 10.1177/2325967118798621. eCollection 2018 Sep. PMID 30263901
- [Background] Mansourvar M, Ismail MA, Raj RG, Kareem SA, Aik S, Gunalan R, Antony CD. The applicability of Greulich and Pyle atlas to assess skeletal age for four ethnic groups. J Forensic Leg Med. 2014 Feb;22:26-9. doi: 10.1016/j.jflm.2013.11.011. Epub 2013 Dec 3. PMID 24485416
- [Background] Iwano T, Kurosawa H, Tokuyama H, Hoshikawa Y. Roentgenographic and clinical findings of patellofemoral osteoarthrosis. With special reference to its relationship to femorotibial osteoarthrosis and etiologic factors. Clin Orthop Relat Res. 1990 Mar;(252):190-7. PMID 2302884
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470